CLINICAL TRIAL: NCT03808935
Title: A Double-Blind, Placebo-Controlled, Parallel-Group Study of Cannabidiol Plus Tetrahydrocannabinol (CBD+THC) Given as Adjunctive Therapy in Patients With Refractory Seizures
Brief Title: Cannabis Extract in Refractory Epilepsy Study
Acronym: CERES
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Participants are no longer being examined or receiving intervention.
Sponsor: The Epilepsy Research Program of the Ontario Brain Institute (Other)
Collaborators: Ontario Brain Institute (Other); University of Toronto (Other); University Health Network, Toronto (Other); London Health Sciences Centre (Other); MedReleaf (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPL29
Record Dates: First submitted 2019-01-11; First posted 2019-01-18 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Drug Resistant Epilepsy
Keywords: epilepsy; drug resistant; refractory; seizures; cannabidiol; cbd; cannabis
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy; Seizures; Color Vision Defects; Marijuana Abuse | interventions — Medical Marijuana

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical cannabis (Experimental): Capsules containing cannabis extract, dissolved in high-oleic sunflower oil, and CBD/THC in a 16:1 ratio.
  Interventions: Drug: Medical Cannabis
- Placebo Control (Placebo Comparator): Capsules containing a high-oleic sunflower oil, calorie-equated to the active treatment. There will be no active compounds in the placebo treatment.
  Following treatment with placebo, all participants in this group will begin treatment with medical cannabis.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Medical Cannabis — The experimental intervention will begin with two weeks of titration (100 mg to 200 mg of CBD per day), followed by four weeks of treatment (maximum 300 mg of CBD per day) and four weeks of maintenance (maximum 300 mg of CBD per day). A two week washout phase will slowly decrease the daily dose (200 mg to 100 mg of CBD per day). All daily doses are equally divided into a morning and evening dose.
  Other Names: CBD/THC
  Arms: Medical cannabis
Drug: Placebo — The placebo intervention will begin with two weeks of titration, followed by four weeks of treatment. Participants will then be unblinded to their study group and begin two weeks of titration, four weeks of treatment, and two weeks of washout with medical cannabis, following the same dosing and schedule as the experimental group. All daily doses are equally divided into a morning and evening dose.
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to examine whether a low dose of CBD+THC will decrease the frequency of convulsive seizures in adults with drug-resistant epilepsy, when used in addition to standard anti-epileptic drugs (AEDs). This study will also study the genes associated with epilepsy and whether different epileptic syndromes respond to treatment with CBD+THC.

DETAILED DESCRIPTION:
Background: Cannabidiol (CBD) and Δ9-tetrahydrocannabinol (THC) are the two major compounds found in the cannabis plant. Reports from patients, families, and the scientific community suggest that CBD (when used as an add-on therapy) decreases the number of convulsive seizures in children and adults with Dravet syndrome, Lennox-Gastaut syndrome, and Tuberous sclerosis complex.

Trial design: Phase III, double-blind, randomized, placebo-controlled, parallel-group trial, followed by an open phase where treatment allocation will be revealed and all participants will either continue or begin receiving the active study drug.

Participants: Adults (18 years of age and older) with drug-resistant epilepsy, including patients with Dravet and Lennox Gastaut syndromes, and patients with frequent convulsive seizures (e.g., tonic, tonic-clonic, atonic, drop attacks, and focal motor seizures).

Interventions: Capsules containing a ratio of 16 CBD: 1 THC oil at a maximum total daily dose of approximately 300 mg of CBD per day, divided into equal doses in the morning and evening.

Comparator: Placebo capsules containing high-oleic sunflower oil and no active or medicinal ingredients.

Outcomes: Frequency of seizures; side effects; blood levels of AEDs, CBD, THC, and liver enzymes; impact on cognition and quality of life; genetics.

Sample size: A total of 80 participants (40 assigned to treatment and 40 to control group) recruited from Toronto Western Hospital in Toronto, and University Hospital in London, Ontario.

Time: Each participant will be enrolled for approximately 16 to 18 weeks, while the clinical trial is expected to take place over a period of two years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy according to the ILAE classification.
* At least 4 motor seizures per month at the start of the study, despite treatment with at least two different anti-epileptic drugs (given concurrently or sequentially) for at least one year.
* At least 4 motor seizures per month during the prospective baseline phase (4 weeks) with no 21-day seizure free periods.
* Stable dose(s) of the same AED(s) for one month prior to screening.
* Agrees not to take any cannabinoids during the study or any other investigational compound for one month before the study or outside cannabinoids during the study.
* Is planning to stay in Canada for the duration of the trial.
* Is able to travel to one of the study sites for in-person visits with the study physicians and to a local lab for blood collection.
* Has access to telephone, computer, and internet for regular correspondence and to complete the study questionnaires.

Exclusion Criteria:

* Participation in a study involving administration of an investigational compound within one month of Visit 1.
* Evidence of clinically significant non-epileptic disease (cardiac, respiratory, gastrointestinal, hepatic, hematologic, or renal disease, etc.) that in the opinion of the investigators could affect the patient's safety or trial conduct.
* Progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
* Occurrence of psychogenic seizures in the previous year.
* History of drug misuse/abuse (other than cannabinoids). Consideration may be given to allowing inclusion of subjects with remote history of drug abuse (within a defined relevant time period).
* Multiple drug allergies (dermatological, hematological, or organ toxicity) or more than one severe drug reaction(s).
* Pregnancy, breastfeeding.
* Known or suspected hypersensitivity to cannabinoids, or any of the excipients of the investigational medicinal product.
* Patients with a history of major depression, suicidal ideation or attempted suicide, schizophrenia or any other psychotic disorder, patients with a family history of schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Frequency of convulsive seizures | 0 - 10 weeks

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by the adverse events questionnaire | 0- 10 weeks
Changes in blood levels of CBD and THC from baseline to end of treatment | 0 - 10 weeks
Changes in blood levels of AEDs from baseline to end of treatment | 0 - 10 weeks
Changes in blood levels of liver enzymes AST, ALT, and GGT from baseline to end of treatment | 0 - 10 weeks
Changes in quality of life from baseline to end of treatment as assessed by the Quality of Life in Epilepsy Inventory (QOLIE-31) questionnaire | 0 - 10 weeks
  QOLIE-31 is a 31-item measure assessing health-related quality of life in adults with epilepsy. Seven scales assess seizure worry, overall quality of life, emotional well-being, cognitive and medication effects, and social function.
Changes in quality of life from baseline to end of treatment as assessed by the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire | 0 - 10 weeks
  WHOQOL-BREF is a 26-item measure of physical health, psychological health, social relationships, and environment.
Changes in quality of life from baseline to end of treatment as assessed by the Quality of Life Childhood Epilepsy (QOLCE) questionnaire | 0 - 10 weeks
  QOLCE is a 55-item scale assessing health-related quality of life in children with epilepsy from the perspective of the parent or caregiver. It covers cognitive, emotional, social, and physical functioning.
Changes in symptoms of depression from baseline to end of treatment as assessed by the Neurological Disorder Depression Inventory for Epilepsy (NDDI-E) | 0 - 10 weeks
  NDDI-E is a 6-item questionnaire designed to screen for depression in adults with epilepsy.
Changes in symptoms of depression from baseline to end of treatment as assessed by the Quick Inventory of Depressive Symptoms (QIDS) | 0 - 10 weeks
  QIDS is a 16-item measure designed to assess the severity of depressive symptoms.
Changes in symptoms of anxiety from baseline to end of treatment as assessed by the Generalized Anxiety Disorder 7-item (GAD-7) | 0 - 10 weeks
  GAD-7 is a 7-item questionnaire assessing severity of generalized anxiety disorder.
Change in overall severity of epilepsy from baseline to end of treatment as assessed by the Global Analysis of Severity of Epilepsy Scale (GASE) | 0 - 10 weeks
  GASE is a single-item, 7-point global rating scale that was designed to assess the overall severity of epilepsy.
Change in quality of sleep from baseline to end of treatment as assessed by the Pittsburgh Sleep Quality Index (PSQI) | 0 - 10 weeks
  PSQI is a 19-item measure assessing subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication and daytime dysfunction.
Change in participant's impression of change from baseline to end of treatment as assessed by the Patients' Global Impression of Change (PGIC) scale | 0 - 10 weeks
  PGIC is a 7-point scale assessing the patient's perspective of overall improvement and efficacy of treatment. Scores range from "very much improved" to "very much worse".
Change in caregiver's impression of change from baseline to end of treatment as assessed by the Caregiver's Global Impression of Change (CGIC) scale | 0 - 10 weeks
  CGIC is a 7-point scale assessing the caregiver's perspective of overall improvement and efficacy of treatment. Scores range from "very much improved" to "very much worse".
Changes in psychological symptoms from baseline to end of treatment as assessed by the Brief Symptom Inventory (BSI-53) | 0 - 10 weeks
  BSI-53 is a 53-item measure assessing psychological profiles. It covers 9 primary domains: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism.
Changes in functional impairment from baseline to end of treatment as assessed by the Sheehan Disability Scale (SDS) | 0 - 10 weeks
  SDS is a 5-item measure assessing functional impairment in three inter-related domains: work/school, social, and family life.

CONTACTS AND LOCATIONS:
Overall Officials: W M Burnham, PhD, Principal Investigator — University of Toronto; Peter Tai, MD, Principal Investigator — University Health Network, Toronto; Seyed Mirsattari, MD, Principal Investigator — London Health Sciences Centre; Nancy Mingo, MD, Principal Investigator — University Health Network, Toronto; Danielle Andrade, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - University Hospital Campus, London Health Sciences Centre, London, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario